CLINICAL TRIAL: NCT02586116
Title: Post Market Comparison of nanOss Cervical Interbody Fusion System to C-Plus Interbody Fusion Device With Autograft
Brief Title: Comparison of nanOss Cervical IBF System to C-Plus PEEK IBF Device With Autograft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI Surgical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NC03
Record Dates: First submitted 2015-10-16; First posted 2015-10-26 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Intervertebral Disc Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- nanOss (Active Comparator): nanOss Cervical IBF System with nanOss BA Bone Void Filler
  Interventions: Device: nanOss
- C-Plus (Active Comparator): C-Plus PEEK IBF Device with autograft
  Interventions: Device: C-Plus

INTERVENTIONS:
Device: nanOss — nanOss Cervical Interbody Fusion Device with nanOss BA bone void filler.
  Other Names: nanOss Cervical IBF Device
  Arms: nanOss
Device: C-Plus — C-Plus PEEK IBF Device with autograft
  Other Names: C-Plus PEEK IBF Device
  Arms: C-Plus

SUMMARY:
This is a post-market, prospective, randomized clinical investigation to evaluate the performance of the nanOss Cervical Interbody Fusion (IBF) device with nanOss Bioactive Bone Void Filler for the treatment of cervical disc disease. A secondary objective is to compare the performance of the nanOss Cervical IBF Device and nanOss Bioactive Bone Void Filler with the performance of the C-Plus PEEK IBF Device with autograft. This study will enroll 40 patients at one (1) site. After subjects have signed an informed consent, they will be randomly assigned to either the nanOss Cervical IBF device arm or the C-Plus PEEK IBF Device. Patients will complete the preoperative visit and examinations. Patients will be evaluated at discharge, six (6) weeks, three (3) months, six (6) months, and twelve (12) months. Patients will be evaluated at twenty-four (24) months post-operatively if they have not demonstrated fusion at the 12 month time point.

DETAILED DESCRIPTION:
The nanOss Cervical Interbody Fusion Device is CE-marked for single level intervertebral body fusion from C3 to T1 for the treatment of cervical disc disease. The nanOss IBF device is designed to be used as one device per level, with graft material and supplemental fixation.

nanOss BABone Void Filler is a resorbable porous calcium phosphate bone void filler for use as a bone graft substitute or bone void filler. It is CE marked for use as a bone void filler in the spine, and it is to be re-hydrated with Bone Marrow Aspirate (BMA) alone, or a mixture of the patient's BMA and autograft.

The C-Plus PEEK IBF Device is indicated for use in skeletally mature adults at one level in the cervical spine, from C3 to T1, for the treatment of cervical disc disease. The device is to be used in patients who have had six weeks of non-operative treatment. Autogenous bone graft is placed within the central cavity of the C-Plus PEEK IBF Device.

The SlimFuse Cervical Plate System components are titanium alloy plates and screws designed to temporarily provide resistance to flexion, extension, lateral bending and axial rotation with strength and stiffness in the cervical spine (C2-C7) in order to promote cervical fusion. The anterior approach should be used when implanting the SlimFuse Cervical Plate System.

The primary goal of this study is to evaluate the outcomes between nanOss Cervical IBF Device and C-Plus PEEK IBF Device. The primary endpoint will be objectively determined via x-rays and CT scan to assess fusion. Secondary endpoints will include subjective patient scores for neck and arm pain and quality of life along with analysis of the proportion of patients who experience a treatment failure.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 21 years of age and skeletally mature.
2. Must have cervical disc disease (defined as neck pain of discogenic origin with degeneration of the disc confirmed by history and radiographic studies) at one level in the cervical spine between C3 to T1.
3. Must have completed a minimum of six weeks of unsuccessful conservative, non- operative care or has the presence of progressive symptoms or signs of nerve root/spinal cord compression in the face of conservative treatment
4. Has pre-operative objective evidence of primary diagnosis confirmed by appropriate imaging studies (AP/LAT/FLX/EXT X-rays & a recent MRI)
5. Is willing and able to comply with all clinical investigation visits and procedures including screening treatment procedures, post-operative management, the follow-up schedule and completion of forms or questionnaires.
6. Is able to understand and sign the informed consent document

Exclusion Criteria:

1. Requires fusion at more than one level
2. Has had prior fusion at the level to be treated.
3. Has a metabolic or systemic bone disorder.
4. Has a disease that significantly inhibits bone healing (i.e., severe osteoporosis, osteomalacia, Paget's disease)
5. Has a systemic or local infection (active or latent)
6. Has acute or chronic infections in the surgical area (i.e., soft tissue infections; inflammatory, bacterial bone disorders, osteomyelitis)
7. chronic use of steroids, other than episodic use or inhaled corticosteroids
8. has any significant general illness (i.e. tested positive for HIV, Hepatitis B or Hepatitis C, has active metastatic cancer of any type, uncontrolled diabetes Type I, dialysis dependent renal failure, symptomatic liver disease)
9. has a mental or physical condition that would limit the ability to comply with study requirements or would preclude accurate evaluation.
10. Is immunocompromised or being treated with immunosuppressive agents (including chemotherapy or radiation treatment).
11. has documented allergies to hydroxyapatite or porcine collagen, PEEK, titanium, titanium alloy or tantalum.
12. currently pregnant, or interested in becoming pregnant during the clinical investigation follow-up
13. is a smoker
14. is a prisoner
15. is currently involved in another drug or device clinical investigation that may confound the clinical investigation data.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Number of patients demonstrating fusion at 12 months post-operatively | 12 months
  Fusion is defined as the presence of bridging bone between adjacent endplates of the involved motion segment, AND ≤ 2º total angular motion from flexion to extension, AND < 1.25 mm translational motion.

SECONDARY OUTCOMES:
Scores on the Neck Disability Index Questionnaire | 12 months
Pain on the Visual Analog Scale | 12 months
Adverse Events | 12 months
  Serious device related adverse events.
Score on the EQ-5D Health Outcomes Survey | 12 months
Disc Height in millimetres | 12 months
Device Migration in millimetres | 12 months
Device Subsidence in millimetres | 12 months
Score on the RAND 36 item questionnaire | 12 months
Proportion of patients with subsequent surgical intervention | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Peuskens, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao Z, Jiang D, Ou Y, Tang K, Luo X, Quan Z. A hollow cylindrical nano-hydroxyapatite/polyamide composite strut for cervical reconstruction after cervical corpectomy. J Clin Neurosci. 2012 Apr;19(4):536-40. doi: 10.1016/j.jocn.2011.05.043. Epub 2012 Feb 3. PMID 22305868
- [Background] Kim SC, Kang SW, Kim SH, Cho KH, Kim SH. Clinical and radiological outcomes of anterior cervical interbody fusion using hydroxyapatite spacer. J Korean Neurosurg Soc. 2009 Oct;46(4):300-4. doi: 10.3340/jkns.2009.46.4.300. Epub 2009 Oct 31. PMID 19893716
- [Background] Ryken TC, Heary RF, Matz PG, Anderson PA, Groff MW, Holly LT, Kaiser MG, Mummaneni PV, Choudhri TF, Vresilovic EJ, Resnick DK; Joint Section on Disorders of the Spine and Peripheral Nerves of the American Association of Neurological Surgeons and Congress of Neurological Surgeons. Techniques for cervical interbody grafting. J Neurosurg Spine. 2009 Aug;11(2):203-20. doi: 10.3171/2009.2.SPINE08723. PMID 19769500